CLINICAL TRIAL: NCT07073053
Title: The Role of Glucagon-Like Peptide-1 Receptor Agonists in Coronary Artery Diseases and Their Potential Mechanisms
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-02-004C
Record Dates: First submitted 2025-06-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Glucagon-Like Peptide-1 Receptor Agonists; Type 2 Diabetes; Coronary Arterial Disease (CAD)
Keywords: Glucagon-Like Peptide-1 Receptor Agonists; type 2 diabetes; coronary arterial disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- semaglutide 1.0mg weekly (Experimental): continue previous standard treatment with add-on semaglutide
  Interventions: Drug: Semaglutide 1.0 mg
- semaglutide 0.5mg weekly (Active Comparator): continue previous standard treatment with add-on semaglutide
  Interventions: Drug: Semaglutide 0.5 mg
- control (No Intervention): continue previous standard treatment

INTERVENTIONS:
Drug: Semaglutide 1.0 mg — add-on current standard treatment which includes SGLT2 inhibitor
  Arms: semaglutide 1.0mg weekly
Drug: Semaglutide 0.5 mg — add-on current standard treatment which includes SGLT2 inhibitor
  Arms: semaglutide 0.5mg weekly

SUMMARY:
The investigators plan to enroll 60 patients from the outpatient clinics or inpatient wards of the Metabolism and Cardiology departments who, within the past three months, have undergone coronary angiography for the treatment of coronary artery disease, are currently using sodium-glucose cotransporter-2 (SGLT-2) inhibitors for glycemic control, and have not received glucagon-like peptide-1 receptor agonist (GLP-1 RA) therapy for more than three months. A randomized controlled clinical trial will be conducted, with 20 participants randomly assigned to receive semaglutide (a GLP-1 RA) at 1 mg once weekly for 6 months, another 20 participants to receive semaglutide at 0.5 mg once weekly for 6 months, and the control group (20 participants) to continue with standard treatment for 6 months. The effects after 6 months will be evaluated in terms of endothelial function, glycemic control indicators including glycemic variability assessed via continuous glucose monitoring (CGM), oxidative stress markers, and the incidence of symptomatic hypoglycemia.

According to the treatment guidelines for type 2 diabetes, either GLP-1 receptor agonists or SGLT-2 inhibitors should be prioritized in patients with type 2 diabetes and coronary artery disease. Therefore, the medication choices in both the intervention and control groups in this study align with current treatment guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. adults (>=20 years old),
2. Type 2 Diabetes with coronary arterial disease underwent angioplasty within 3 months with SGLT2 inhibitors -

Exclusion Criteria:

1. age<20 years old,
2. pregnant women,
3. eGFR<30 ml/min/1.73m2,
4. received GLP-1 agonist in the recent 3 months -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
change of Time-in-range (%) | From enrollment to the end of treatment at 24 weeks
  continuous glucose monitor, time-in-range defined as percentage of time in range of 70-180 blood glucose levels. Change of time-in-range means time-in-range at week 24 - time-in-range at baseline.
change of HbA1c | From enrollment to the end of treatment at 24 weeks
  HbA1c at week 24 - HbA1c at baseline
change of Flow-Mediated Dilatation (FMD) | From enrollment to the end of treatment at 24 weeks
  Flow-Mediated Dilatation (FMD) at week 24 - Flow-Mediated Dilatation (FMD) at baseline

SECONDARY OUTCOMES:
change of serum ROS measurements | From enrollment to the end of treatment at 24 weeks
  serum ROS measurements at week 24 - serum ROS measurements at baseline
change of Peripheral Arterial Tonometry (PAT) | From enrollment to the end of treatment at 24 weeks
  Peripheral Arterial Tonometry (PAT) at week 24 - Peripheral Arterial Tonometry (PAT) at baseline
Hypoglycemic episodes | from enrollment to the end of treatment at week 24.
  the amount of hypoglycemic episodes during the treatment period of 24 weeks. hypoglycemic episodes defined as blood sugar levels less than 50 or with hypoglycemic symptoms.
change of fasting glucose | From enrollment to the end of treatment at week 24
  fasting glucose ar week 24 - fasting glucose at baseline

OTHER OUTCOMES:
change of serum IL-1β | From enrollment to the end of treatment at 24 weeks
  levels of serum IL-1β at week 24 - levels of serum IL-1β at baseline
change of serum IL-6 | From enrollment to the end of treatment at 24 weeks
  levels of serum IL-6 at week 24 - levels of serum IL-6 at baseline
change of serum IL-10 | From enrollment to the end of treatment at 24 weeks
  levels of serum IL-10 at week 24 - levels of serum IL-10 at baseline
change of serum TNF-α | From enrollment to the end of treatment at 24 weeks
  levels of serum TNF-α at week 24 - levels of serum TNF-α at baseline
change of urinary 8-iso PGF 2alfa | From enrollment to the end of treatment at 24 weeks
  urinary 8-iso PGF 2alfa at week 24 - urinary 8-iso PGF 2alfa at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The IPD share plan was not mentioned in this patient consent form.